CLINICAL TRIAL: NCT03702439
Title: Prostate Cancer Screening Trial Using A Group of Radiological Approaches Including MRI and Ultrasound
Brief Title: Prostate Cancer Screening Trial Using Imaging
Acronym: PROSTAGRAM
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18HH4595
Record Dates: First submitted 2018-10-02; First posted 2018-10-11 (Actual); Results first posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Prostate Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participants will be recruited from the community and attend a screening clinic and undergo the following screening tests:

1. Bi-parametric MRI - reported by a radiologist and CAD-AI system
2. Multiparametric ultrasound - including shearwave elastography
3. A standard-of-care PSA test

A systematic +/- targeted biopsy will be performed if any tests are positive, independent of the other tests.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged between 50 and 69 years inclusive at the time of study entry
2. Participants must be fit to undergo all procedures listed in the protocol
3. Estimated life expectancy of 10 years or more
4. An understanding of the English language sufficient to understand written and verbal information about the trial and consent process
5. Participants must be willing and able to provide written informed consent

Exclusion Criteria:

1. Previous PSA test or prostate MRI within the prior two years of screening/consent visit
2. Evidence of a urinary tract infection or history of acute prostatitis within the last 6 months
3. Previous history of prostate cancer, prostate biopsy or treatment for prostate cancer
4. Any potential contraindication to MRI
5. Any potential contraindication to prostate biopsy
6. Dementia or altered mental status that would prohibit the understanding or rendering of informed consent.
7. Any other medical condition precluding procedures described in the protocol

Ages: 50 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men aged 50-69 years
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AHMED HASHIM, Prof, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eldred-Evans D, Winkler M, Klimowska-Nassar N, Burak P, Connor MJ, Fiorentino F, Day E, Price D, Gammon M, Tam H, Sokhi H, Padhani AR, Ahmed HU. Perceived patient burden and acceptability of MRI in comparison to PSA and ultrasound: results from the IP1-PROSTAGRAM study. Prostate Cancer Prostatic Dis. 2023 Sep;26(3):531-537. doi: 10.1038/s41391-023-00662-6. Epub 2023 Mar 31. PMID 37002379
- [Derived] Wurnschimmel C, Kachanov M, Wenzel M, Mandel P, Karakiewicz PI, Maurer T, Steuber T, Tilki D, Graefen M, Budaus L. Twenty-year trends in prostate cancer stage and grade migration in a large contemporary german radical prostatectomy cohort. Prostate. 2021 Sep;81(12):849-856. doi: 10.1002/pros.24181. Epub 2021 Jun 10. PMID 34110033

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant enrollment (411) exceeded the planned protocol enrollment (406) due to the logistics of mpMRI at the screening site. The TMG agreed that over-recruitment could occur on a single day to maximize MRI availability
Groups:
- MRI, PSA and US Group: Men eligible for screening with a short MRI or PSA or ultrasound
Period: Overall Study
Arm/Group | MRI, PSA and US Group
Started | 408
Completed | 408
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Includes men consented and eligible for all screening test
Groups:
- MRI, PSA and US Group: Men screened by PSA, MRI and US
Arm/Group | MRI, PSA and US Group
Number analyzed (Participants) | 408
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 352
  >=65 years | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 408
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 94
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 132
  White | 155
  More than one race | 9
  Unknown or Not Reported | 18

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Men With a Positive MRI Defined by a Score of 3 or Greater
Description: Men with a positive MRI defined by a score of 3 or greater
Time Frame: Through study completion, an average of 1 month
Population: All patients who had an MRI screening test
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Short MRI Arm: Men who had a Short MRI in study
Arm/Group | Short MRI Arm
Number analyzed (Participants) | 406
Percentage of participants | 17.7 [14.3 to 21.8]

2. Secondary Outcome: The Proportion of Men With Screen-positive Prostate MRI Defined by a Score of 4 or Greater
Description: Men With Screen-positive Prostate MRI Defined by a Score of 4 or Greater
Time Frame: Through study completion, an average of 1 month
Population: All men who had a short MRI
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Short MRI Arm
Number analyzed (Participants) | 406
Percentage of participants | 10.6 [7.9 to 14]

3. Secondary Outcome: The Proportion of Men With Screen-positive Prostate US Defined by a Score of 3 or Greater
Description: Men With Screen-positive Prostate US Defined by a Score of 3 or Greater
Time Frame: Through study completion, an average of 1 month
Population: All men who had a ultrasound
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Ultrasound Arm: Men who had a ultrasound in study
Arm/Group | Ultrasound Arm
Number analyzed (Participants) | 405
Percentage of participants | 23.7 [19.8 to 28.1]

4. Secondary Outcome: The Proportion of Men With Screen-positive Prostate US Defined by a Score of 4 or Greater
Description: Men With Screen-positive Prostate US Defined by a Score of 4 or Greater
Time Frame: Through study completion, an average of 1 month
Population: All men who had a ultrasound
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ultrasound Arm
Number analyzed (Participants) | 405
Percentage of participants | 12.8 [9 to 16.5]

5. Secondary Outcome: The Proportion of Men With Screen-positive PSA Defined by a >/=3ng/ml
Description: Men with screen-positive PSA defined by a >/=3ng/ml
Time Frame: Through study completion, an average of 1 month
Population: Men with screen-positive PSA defined by a >/=3ng/ml
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- PSA Arm: Men who had a PSA and one other screening test
Arm/Group | PSA Arm
Number analyzed (Participants) | 406
Percentage of participants | 9.9 [7.3 to 13.2]

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were recorded and monitored continuously until the last study visit, an average of 1.5 months
Arm/Group | MRI, PSA and US Group
All-Cause Mortality (participants affected / at risk) | 0/408
Serious Adverse Events (participants affected / at risk) | 0/408
Other Adverse Events (participants affected / at risk) | 0/408

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT03702439/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT03702439/SAP_001.pdf